CLINICAL TRIAL: NCT00418951
Title: Open, Randomized Comparative Trial of Two Different Schedules of Liposomal Amphotericin B Versus Oral Voriconazole for the Prevention of Invasive Fungal Infections
Brief Title: Liposomal Amphotericin B (Ambisome) Versus Oral Voriconazole for the Prevention of Invasive Fungal Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006-0536
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Results first posted 2011-05-13 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: Voriconazole; Vfend; Liposomal amphotericin B; Ambisome; Acute Myelogenous Leukemia; Myelodysplastic Syndrome; AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Voriconazole; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Liposomal amphotericin B: 3 mg/kg (Experimental): 3 mg/kg intravenously (IV) three times per week
  Interventions: Drug: Liposomal amphotericin B
- Liposomal amphotericin B: 9 mg/kg (Experimental): 9 mg/kg IV once per week
  Interventions: Drug: Liposomal amphotericin B
- Voriconazole: 400 mg (Experimental): 400 mg oral twice daily day 1 followed by 200 mg twice daily
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — 400 mg by mouth twice daily on day 1, followed by 200 mg by mouth twice daily
  Other Names: Vfend
  Arms: Voriconazole: 400 mg
Drug: Liposomal amphotericin B — 3 mg/kg intravenously three times per week over 2 hours +/- 15 minutes
  Other Names: Ambisome
  Arms: Liposomal amphotericin B: 3 mg/kg
Drug: Liposomal amphotericin B — 9 mg/kg intravenously once per week over 2 hours +/- 15 minutes
  Other Names: Ambisome
  Arms: Liposomal amphotericin B: 9 mg/kg

SUMMARY:
The goal of this clinical research study is to compare the effectiveness of liposomal amphotericin B given three times per week , versus liposomal amphotericin B given once per week, versus oral voriconazole in the prevention of fungal infections in patients with acute myeloid leukemia (AML) or myelodysplastic syndromes MDS who are receiving chemotherapy. The safety of these treatments will also be studied and compared.

DETAILED DESCRIPTION:
Ambisome and voriconazole are drugs that have been used to fight fungal infections, which typically occur during chemotherapy as a result of lowered immune system functioning. Ambisome works by binding to the sterol component of the fungal cell membrane. This causes "holes" to appear in the membrane, which leads to death of the fungal cell. Voriconazole inhibits an essential step of the biosynthesis of an important component of the fungal cell wall (ergosterol). This causes the impairment of the fungal cell wall.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will be asked questions about your medical history. You will have a complete physical exam and a chest x-ray. You will have computed tomography (CT) scans of the chest. You will also have about 1 teaspoon of blood drawn for routine tests. Test results from the pregnancy test that you will have before your leukemia treatment will be looked at for this study. You will not have a pregnancy test performed for this study.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to one of 3 treatment groups (Group 1, Group 2, or Group 3). Participants in Groups 1 and 2 will receive treatment with ambisome. Participants in Group 3 will receive treatment with voriconazole. Participants in all 3 groups will begin treatment 24 hours after the last dose of chemotherapy.

If you are assigned to Group 1, you will receive ambisome by vein as a continuous infusion over 2 hours 1 time per day, 3 times each week.

If you are assigned to Group 2, you will receive ambisome by vein as a continuous infusion over 2 hours 1 time per week.

If you are assigned to Group 3, you will take 2 pills by mouth (1 hour after breakfast) and 2 pills by mouth (1 hour after dinner) for 1 day, which amounts to 4 pills in total on Day 1. You will then take 1 pill by mouth (1 hour after breakfast) and 1 pill by mouth (1 hour after dinner) everyday for the remainder of this study, which amounts to 2 pills in total each day.

You will have about 1 teaspoon of blood drawn for routine tests 2 times each week. You will also receive treatment with standard of care medications. These medications (which will be specified by your doctor) will be used to help decrease the risk of developing bacterial infections and viral infections.

If you develop a fever during treatment on this study, you will have a chest x-ray and a CT scan of the chest within 3 days after the fever started.

You may remain on this study for up to 35 days (if you are receiving chemotherapy for the first time) and up to 42 days (if you have had prior chemotherapy). Your participation may end on this study if your study doctor thinks it is necessary, if other antifungal therapy is required, or if you develop any intolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML or high risk MDS undergoing induction chemotherapy or first salvage chemotherapy.
* Age >/=18 years.
* Patients must sign an informed consent.

Exclusion Criteria:

* Patients with history of anaphylaxis attributed to azole or amphotericin B compounds.
* Patients with clinical or other evidence that indicates that they have proven or probable invasive fungal infection prior to enrollment.
* Patients with total bilirubin levels > 3 times the upper normal limits (i.e. > 3.0 mg/dl); or serum glutamic pyruvic transaminase (SGPT)> 5 times upper limit normal.
* Patients with serum creatinine > 2.0 mg/dl.
* Patients receiving any medication that is contraindicated with the use of voriconazole.
* Patients who have participated in this study during induction chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria N Mattiuzzi, MD, Principal Investigator — M.D. Anderson Cancer Center; Gloria N Mattiuzzi, MD, Study Director — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 11/3/2006 to 8/4/09. All patients registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Eight of 120 patients registered never received study drug, therefore were excluded from the study.
Period: Overall Study
Arm/Group | Liposomal Amphotericin B: 3 mg/kg | Liposomal Amphotericin B: 9 mg/kg | Voriconazole: 400 mg
Started | 39 | 33 | 40
Completed | 39 | 33 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Amphotericin B: 3 mg/kg | Liposomal Amphotericin B: 9 mg/kg | Voriconazole: 400 mg | Total
Number analyzed (Participants) | 39 | 33 | 40 | 112
Age Continuous [Median (Full Range); unit: years] | 60 [25 to 84] | 71 [23 to 78] | 71 [19 to 80] | 60 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 19 | 54
  Male | 20 | 17 | 21 | 58
Region of Enrollment [Number; unit: participants]
  United States | 39 | 33 | 40 | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Invasive Fungal Infection
Description: Endpoint was whether participant had an invasive fungal infection or not, a potentially fatal complication with leukemia patients. Efficacy defined as absence of proven and probable fungal infection. Probable fungal infection is: 1) Positive radiographic findings consistent with fungal infections documented on CT imaging: Lower respiratory tract infection: halo sign, air crescent-sign, or cavity within areas of consolidation; Sinus: erosion of sinus walls or extension of infection to neighboring structures, extensive skull base destruction; and/or 2) Two positive galactomannan index test.
Time Frame: 35 days from the start of therapy for induction participants and 42 days for salvage participants.
Population: Outcome evaluability required at least two doses of study drug.
Measure: Number; unit: participants
Arm/Group | Liposomal Amphotericin B: 3 mg/kg | Liposomal Amphotericin B: 9 mg/kg | Voriconazole: 400 mg
Number analyzed (Participants) | 35 | 28 | 39
participants | 3 | 4 | 2

ADVERSE EVENTS:
Time Frame: Three years, ten months.
Arm/Group | Liposomal Amphotericin B: 3 mg/kg | Liposomal Amphotericin B: 9 mg/kg | Voriconazole: 400 mg
Serious Adverse Events (participants affected / at risk) | 5/39 | 2/33 | 4/40
Other Adverse Events (participants affected / at risk) | 0/39 | 0/33 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Amphotericin B: 3 mg/kg (N=39) | Liposomal Amphotericin B: 9 mg/kg (N=33) | Voriconazole: 400 mg (N=40)
Supravnetricular Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0) | 2 (2) — unrelated to study drug
Allergic Reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infection Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Elevated alanine aminotransferase (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes